CLINICAL TRIAL: NCT02204774
Title: Is Obstructive Sleep Apnoea a Risk Factor for Thoracic Aortic Aneurysm Expansion? A Prospective Cohort Study.
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Malcolm Kohler, Head, Division of Pneumology, University of Zurich
Other Study IDs: V 1.1; NCT02162108 (obsolete NCT alias)
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Aortic Aneurysm; Obstructive Sleep Apnea
Keywords: aortic aneurysm; obstructive sleep apnea
MeSH Terms: conditions — Aortic Aneurysm; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dilatated or aneurysmatic Aorta: Complete cohort, which will be followed over 3 years

SUMMARY:
The objective of this prospective cohort study in patients with a known thoracic aortic aneurysm is to test the hypothesis that yearly aneurysm progression rate is higher in patients with obstructive sleep apnoea (OSA) compared to patients without OSA, and that the need for aortic operation or proven or presumed death from aortic rupture or dissection happens more often in patients with thoracic aortic aneurysm and OSA compared to patients without OSA.

DETAILED DESCRIPTION:
Thoracic aortic aneurysm An aortic aneurysm is defined as a localised dilatation of the aorta, which includes all three layers of the vessel, intima, media and adventitia. The incidence of thoracic aortic aneurysm is estimated to be six to ten cases per 100,000 patient years, most commonly occurring in the sixth and seventh decade of life. Thoracic aortic aneurysms are two to four times more commonly found in males than in females. Sixty percent of thoracic aortic aneurysms involve the ascending aorta, 40% the descending aorta, and 10% involve the thoraco-abdominal aorta. The pathogenesis and natural history as well as the therapy of thoracic aortic aneurysms differ for each of these segments.

Thoracic aneurysms of the ascending aorta are considered to result from cystic degeneration of the media layer, a process associated with weakening of the aortic wall. Cystic medial degeneration occurs with aging, but seems to be increased in some families and with arterial hypertension. Other risk factors which have been suggested to be associated primarily with thoracic aneurysm formation of the descending aorta are the same as those for atherosclerosis (e.g. hypertension, smoking and hypercholesterolemia). Whether atherosclerosis itself is a prerequisite for aortic aneurysm development is a matter of debate. A multifactorial, non-atherosclerotic cause such as a defect in vascular structural proteins and breakdown of extracellular matrix proteins in combination with increased mechanical stress has been postulated as the most likely mechanism for thoracic aneurysm formation.

Transthoracic echocardiography, computed tomography or MR angiography are recommended for serial re-evaluation of a thoracic aortic aneurysm.

Natural history data on thoracic aortic aneurysms is scarce; however, aneurysm diameter has been shown to increase by 1 to 10 mm per year. The rate of expansion is related to the diameter of the aneurysm with larger aneurysms expanding faster; the findings of an early cohort study on the natural course of thoracic aortic aneurysms found a yearly expansion of 7.9mm in aneurysms >50mm, compared to 1.7mm in aneurysms ≤50mm.

In several series of patients, aneurysm rupture occurred in 32% to 68% of medically treated patients. The most important identified risk factor for rupture seems to be the size of the aneurysm; the yearly rate of dissection or rupture ranges from 2%, to 3%, to 7%, for thoracic aortic aneurysms less than 50 mm, 50-59 mm, and ≥60 mm in diameter, respectively. Expansion rate per year, male gender, hypertension, systemic steroid therapy and inflammation are other factors associated with increased risk of aneurysm rupture.

Asymptomatic patients with a thoracic aortic aneurysm are usually managed medically with blood pressure control using a beta blocker and serial evaluation of aneurysmal size progression. Surgery is reserved for symptomatic patients, and for asymptomatic patients with rapid aneurysm expansion (usually defined as >10mm per year), or an aneurysm diameter >50 to 60mm, depending on the affected aortic segment, body size and other clinical factors. However, thoracic aneurysm repair is associated with high morbidity and mortality rates between 3% and 12% in more recent retrospective series. In cases of emergency surgery for thoraco-abdominal aneurysm the 30 day mortality has even been reported to be as high as 40%.

Therefore, any modifiable factors influencing the onset of a thoracic aneurysm and its progressive expansion are of major interest, hopefully leading to new therapeutic strategies to improve morbidity and mortality.

Obstructive sleep apnoea (OSA) is characterised by a repetitive collapse of the pharynx during sleep, which results in apnoea or hypopnoea associated with oxygen desaturations and arousals from sleep, often many hundred times per night. OSA, defined as apnoea-hypopnoea index (AHI) of 5/h or higher, is a common but underdiagnosed sleep-related breathing disorder affecting up to 25% of the middle-aged male population twenty years ago, that now is substantially increased due to higher prevalence of obesity. It is estimated that 80-90% of moderate to severe OSA are not diagnosed. The gold-standard diagnostic test for OSA is in-laboratory polysomnography. Alternatively, OSA can be diagnosed with high sensitivity and specificity - in subjects with high probability for OSA based on clinical symptoms - by in-hospital respiratory polygraphy or portable monitor devices at home (cardiorespiratory sleep study). The usual and most effective treatment for OSA is continuous positive airway pressure (CPAP) therapy. A device delivers a continuous level of positive airway pressure with fixed or auto-titrating pressure keeping airway patency and thereby preventing apnoeas and hypopnoeas.

Preliminary data from observational and non-randomised studies indicate an association between OSA and cardiovascular events. There is also evidence that severe symptomatic sleep apnoea is associated with hypertension, stroke and myocardial infarction. The proposed mechanisms underpinning the association between OSA and vascular dysfunction leading to cardio- and cerebrovascular disease are increasingly large intrathoracic pressure changes leading to mechanical stress on the heart and large artery walls, arousal-induced reflex sympathetic activation with resultant repetitive blood pressure rises, sometimes to over 200mmHg, and intermittent hypoxia leading to increased oxidative stress and sympathetic activity. The rises in blood pressure induce extensive shear stresses on blood vessel walls - forces that are thought to cause vascular wall damage.

Recent findings from observational studies suggest a possible link between OSA, thoracic aortic dilatation and aortic events in patients with Marfan's syndrome. Marfan's syndrome is an inherited disorder of the connective tissue and aortic root dilatation with subsequent rupture is the commonest life-threatening manifestation. In a cross-sectional study including patients with Marfan's syndrome, the severity of OSA was positively correlated with the diameter of the aortic root. In a recent prospective Marfan cohort study, the rate of aortic events (defined as operation because of rapid progressive aortic dilatation, and death because of aortic rupture) was compared between patients with and without OSA. Aortic-event free survival was significantly shorter in patients with Marfan's syndrome and OSA compared to patients without OSA, suggesting that OSA may be an important risk factor for aortic events in Marfan's syndrome.

The underlying mechanisms through which OSA may promote aortic dilatation are not clear. OSA has been shown to be associated with increased diurnal blood pressure as well as with large and recurrent surges in blood pressure during apnoeic events, which is the main identified risk factor for aortic dilatation and dissection. In addition, obstructive apnoeas are associated with repeated inspiratory effort against the collapsed upper airway causing recurrent large negative intrathoracic pressures (sometimes as low as -80 mmHg) and thereby producing outward radial forces on intrathoracic structures including the aorta. This hypothesis is supported by the findings of Peters et al. who reported increased aortic diameters during obstructive apnoeas in an animal model. In healthy humans, experimentally simulated obstructive apnoea/hypopnoea has also been shown to lead to an acute increase in proximal aortic diameter and transmural pressures.

In a recently published cohort study of patients with abdominal aortic aneurysms, it was shown that severe OSA may be associated with an accelerated expansion of abdominal aortic aneurysms. Because there is only limited cross-sectional and inconclusive data on the possible association between OSA and thoracic aortic aneurysm from non-Marfan study populations a prospective large cohort study of patients with thoracic aortic aneurysms is needed to investigate whether OSA is associated with faster progression of aortic dilatation, and aortic events, in a high risk population. Should OSA appear to be a factor associated with an increased risk for rapid aortic dilatation and aortic events, then a randomised controlled trial in those with OSA would be appropriate, looking at the effect of continuous positive airway pressure (the definitive treatment for OSA) on thoracic aortic dilatation.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of thoracic aortic aneurysm defined by the following parameters

   * Women: at the level of the sinus of valsalva >39mm, or ascending aorta >42mm.
   * Men: at the level of the sinus of valsalva >44mm, or ascending aorta >46mm.
2. Age > 18 years.

Exclusion Criteria:

1. Patients on continuous positive airway pressure (CPAP) therapy for OSA at baseline.
2. Patients with known central sleep apnoea.
3. Patients on morphine or other opioid medication, heroin addiction, alcohol addiction.
4. Patients with moderate or severe aortic regurgitation.
5. Patients with moderate or severe aortic stenosis.
6. Pregnant patients.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of thoracic aortic aneurysm defined by the following parameters
  * Women: at the level of the sinus of valsalva >39mm, or ascending aorta >42mm.
  * Men: at the level of the sinus of valsalva >44mm, or ascending aorta >46mm.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2014-07-05 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Aneurysm expansion rate | three years
  mm per year

SECONDARY OUTCOMES:
combined endpoint of operation (or fulfilling the criteria for operation) | three years
  Operation
endovascular repair because of rapid progression of thoracic aortic aneurysm | three years
  >10 mm per year and/or an aneurysm diameter >50 to 60 mm
Death from proven or presumed aortic dissection/rupture | three years
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, MD, Study Director — Universuty of Zurich
Locations (1):
- University Hospital Zurich, Pneumology, Zurich, Switzerland

REFERENCES:
- [Derived] Gaisl T, Rejmer P, Roeder M, Baumgartner P, Sievi NA, Siegfried S, Stampfli SF, Thurnheer R, Stradling JR, Tanner FC, Kohler M. Obstructive sleep apnoea and the progression of thoracic aortic aneurysm: a prospective cohort study. Eur Respir J. 2021 May 6;57(5):2003322. doi: 10.1183/13993003.03322-2020. Print 2021 May. PMID 33214207